CLINICAL TRIAL: NCT06790888
Title: A Multicenter, Randomized Controlled, Open-Label Study of Ripertamab Combined With Eltrombopag Versus Eltrombopag for ITP Patients After First-Line Steroid Therapy
Brief Title: Ripertamab Plus Eltrombopag vs. Eltrombopag in ITP Patients Post-Steroid Failure
Acronym: RPE-ITP
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Union Hospital, Tongji Medical College, Huazhong University of Science and Technology (Other)
Collaborators: Sinocelltech Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: UHCT240527
Record Dates: First submitted 2024-12-15; First posted 2025-01-24 (Actual); Last update posted 2025-01-24 (Actual); Status verified 2024-11

CONDITIONS: ITP - Immune Thrombocytopenia
Keywords: Ripertamab
MeSH Terms: conditions — Purpura, Thrombocytopenic, Idiopathic | interventions — eltrombopag

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Eltrombopag/Ripertamab (Experimental): Eltrombopag (starting at 2.5mg once daily, 28 days, adjusted based on platelet count),Ripertamab (375 mg/m² BSA on Day 1)，If the participant remains in remission at the 3-month, an additional intravenous dose of 375 mg/m² BSA Ripertamab is administered
  Interventions: Combination Product: Ripertamab/Eltrombopag
- Eltrombopag (Active Comparator): Eltrombopag (starting at 2.5mg once daily, 28 days, adjusted based on platelet count)
  Interventions: Drug: Eltrombopag

INTERVENTIONS:
Combination Product: Ripertamab/Eltrombopag — Ripertamab, a novel anti-CD20 monoclonal antibody, in combination with Eltrombopag . Ripertamab is administered intravenously at a dose of 375 mg/m² BSA on Day 1 . If the participant remains in remission at the 3-month mark, an additional intravenous dose of 375 mg/m² Ripertamab is administered. Eltrombopag are given orally at an initial dose of 2.5 mg once daily, with dosage adjustments made every two weeks based on platelet count response, for a total treatment duration of up to Day 28.
  Other Names: Anti-CD20/TPO-RA
  Arms: Eltrombopag/Ripertamab
Drug: Eltrombopag — Eltrombopag as a single therapy. Eltrombopag is a thrombopoietin receptor agonist given orally at an initial dose of 2.5 mg once daily, with dosage adjustments made every two weeks based on platelet count response, for a total treatment duration of up to Day 28.
  Other Names: TPO-RA
  Arms: Eltrombopag

SUMMARY:
This study aims to evaluate the efficacy and safety of Ripertamab in combination with Eltrombopag compared to Eltrombopag alone for patients with Primary Immune Thrombocytopenia (ITP) who have not responded to or have relapsed after first-line steroid therapy. Participants will be randomly assigned to one of two treatment groups and followed for 52 weeks to assess response rates and safety.

DETAILED DESCRIPTION:
This is a multicenter, open-label, randomized controlled clinical trial designed to compare the effects of Ripertamab plus Eltrombopag versus Eltrombopag monotherapy in adults with ITP. The study will enroll approximately 78 participants, aged 18 to 80 years, who have had an inadequate response to or relapsed after first-line steroid therapy. The primary outcome measure is the sustained response rate at 12 weeks post-treatment initiation. Secondary outcomes include overall response rate, complete response rate, median time to response, median sustained response time, and safety. Participants will undergo regular blood tests and clinical assessments throughout the study period.

ELIGIBILITY:
Inclusion Criteria:

1. Diagnosis: Confirmed Primary Immune Thrombocytopenia (ITP) with an age range of 18 to 80 years, inclusive, and no gender restrictions.
2. Bone Marrow Cytology: Diagnosis via bone marrow cytology excluding secondary thrombocytopenia caused by other diseases, with primary ITP patients who are unresponsive to or have relapsed after first-line steroid therapy (platelet count drops below 30×10^9/L).
3. Coagulation Status: Laboratory tests show prothrombin time (PT/INR) and activated partial thromboplastin time (APTT) not exceeding 20% above the upper limit of normal values, with no history of coagulation disorders other than ITP.
4. Bone Marrow Function: Normal bone marrow function indicated by an absolute neutrophil count (ANC) ≥1.5×10^9/L and hemoglobin (Hb) ≥90 g/L.

Liver and Kidney Function: Normal liver and kidney function with serum direct bilirubin and indirect bilirubin ≤1.5 times the upper limit of normal (ULN); 5.alanine aminotransferase (ALT) and aspartate aminotransferase (AST) ≤3 times the upper limit of normal (ULN); serum creatinine ≤1.5 times the upper limit of normal (ULN).

6.Psychiatric History: No history of psychiatric disorders. 7.Informed Consent: Voluntary signing of an informed consent form.

Exclusion Criteria:

1. Life-Threatening Bleeding: Presence of bleeding that poses an immediate threat to life, such as severe anemia or central nervous system bleeding.
2. Recent Treatment: Use of intravenous immunoglobulin, thrombopoietin receptor agonists, recombinant human thrombopoietin (rhTPO), immunosuppressants, anti-CD20 monoclonal antibodies, or systemic corticosteroids within 28 days prior to enrollment.
3. Malignancy History: History of malignancy.
4. Cardiac Conditions: Presence of severe heart failure or other diseases significantly impacting cardiac function (e.g., unstable angina, congestive heart failure, uncontrolled hypertension, arrhythmias, or prolonged QTc interval within the last 3 months).
5. Coagulation Disorders: History of coagulation disorders other than ITP, such as disseminated intravascular coagulation (DIC), hemolytic uremic syndrome (HUS), or thrombotic thrombocytopenic purpura (TTPP).
6. Viral Markers: Hepatitis C virus (HCV) antibody positive with HCV RNA quantitative test ≥10^4 copies/mL; or Hepatitis B virus (HBV) markers positive for HBsAg and/or HBcAb with HBV DNA positivity.
7. Immunocompromised: History of immunodeficiency, including HIV positivity or other acquired or congenital immunodeficiency diseases, autoimmune diseases, or a history of organ transplantation.
8. Tuberculosis: Suspected active or latent tuberculosis.
9. Active Infections: Presence of active infections at enrollment, or any significant infectious events within 4 weeks prior to enrollment or major surgery within 4 weeks.
10. Pregnancy and Lactation: Pregnant or nursing women, or women of childbearing potential or considering pregnancy during the study period.
11. Other Conditions: Any other conditions deemed by the investigator as contraindications for study participation.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 78 (Estimated)
Dates: Start 2025-02 (Estimated); Primary Completion 2027-12 (Estimated); Study Completion 2027-12 (Estimated)

PRIMARY OUTCOMES:
Sustained Response Rate at 12 Weeks | up to 12weeks
  The primary outcome measure is the proportion of patients who achieve a sustained response at 12 weeks after the initiation of treatment. A sustained response is defined as a platelet count of ≥30×10^9/L without bleeding and without the need for rescue therapy.

SECONDARY OUTCOMES:
Overall Response Rate (ORR) | through study completion, an average of 1 year
  The percentage of patients who achieve any response (complete or partial) to the treatment as measured by an increase in platelet count from baseline.
Complete Response Rate (CR%) | through study completion, an average of 1 year
  The proportion of patients who achieve a complete response, defined as a platelet count of ≥100×10^9/L without bleeding and without the need for rescue therapy.
Median Time to Response (mTTR) | 1 year
  The time at which 50% of the patients achieve a response, measured from the start of treatment until the first evidence of therapeutic effect.
Median Sustained Response Time (mSRT) | 1 year
  The time at which 50% of the patients maintain a response without relapse, measured from the start of treatment until the response is no longer sustained.
24-week Sustained Response Rate (24-week SR) | up to 24 weeks
  The proportion of patients who maintain a sustained response at 24 weeks post-treatment initiation, defined by a platelet count of ≥100×10^9/L without bleeding and without rescue therapy.
52-week Sustained Response Rate (52-week SR) | up to 52 weeks
  The percentage of patients who continue to show a sustained response at 52 weeks after starting treatment, with platelet counts meeting predefined criteria.

CONTACTS AND LOCATIONS:
Overall Officials: Heng MEI, Ph.D&M.D, Study Chair — Union Hospital, Tongji Medical College, Huazhong University of Science and Technology

IPD SHARING:
Plan to Share IPD: No